CLINICAL TRIAL: NCT05244837
Title: Predictive Biomarker for the Efficacy and Safety of the Combination of Chemotherapy and Tislelizumab in Non Small Cell Lung Cancer：a Multicentre Prospective Clinical Trial
Brief Title: Predictive Biomarker for Efficacy and Safety of Combination of Chemotherapy and Tislelizumab in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hao Long (Other)
Responsible Party: Sponsor-Investigator, Hao Long, Chief Physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2020-008
Record Dates: First submitted 2021-10-31; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Tislelizumab; Safety; Biomarker; Chemotherapy
MeSH Terms: interventions — tislelizumab; Carboplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: This study consists includes two groups, one is the treatment of patients with resectable lung cancer and the other is the treatment of patients with unresectable lung cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A:Resectable Stage IIB-IIIA Non Small Cell Lung Cancer (NSCLC) (Experimental): Patients received neoadjuvant treatment with Platinum-based doublet chemotherapy plus tislelizumab(200 mg) on day 1 of each 21-day cycle, for 3-4 cycles before surgical resection, followed by adjuvant intravenous tislelizumab monotherapy for 1 year ( 200 mg every 3 weeks for 2 cycles, followed by 200 mg every 4 weeks for 12 cycles).
  Interventions: Drug: Tislelizumab 200 mg; Drug: Carboplatin AUC 5; Drug: pemetrexed 500mg/m2; Drug: Paclitaxel 175mg/m2; Drug: Nab-paclitaxel 260 mg/m2
- Arm B：Unresectable Stage IIIA/IIIB/IIIC or IV Non Small Cell Lung Cancer (NSCLC) (Experimental): Patients received neoadjuvant treatment with Platinum-based doublet chemotherapy plus tislelizumab(200 mg) on day 1 of each 21-day cycle, for 4-6 cycles , followed by adjuvant intravenous tislelizumab monotherapy ( 200 mg every 3 weeks )，until disease progression or intolerable toxicity If surgery is not possible；If surgery is possible after assessment, subsequent treatment at the discretion of the investigator
  Interventions: Drug: Tislelizumab 200 mg; Drug: Carboplatin AUC 5; Drug: pemetrexed 500mg/m2; Drug: Paclitaxel 175mg/m2; Drug: Nab-paclitaxel 260 mg/m2

INTERVENTIONS:
Drug: Tislelizumab 200 mg — Tislelizumab 200mg IV Q3W + Followed by adjuvant treatment for 1 year (Tislelizumab 200 mg IV Q3W for 2 cycles and Tislelizumab 200 mg Q4W for 12 cycles)
  Other Names: Tislelizumab
Drug: Carboplatin AUC 5 — Carboplatin AUC 5 IV Q3W
  Other Names: Carboplatin
Drug: pemetrexed 500mg/m2 — Pemetrexed 500mg/m2 IV Q3W if non-squamous lung cancer
  Other Names: pemetrexed
Drug: Paclitaxel 175mg/m2 — Paclitaxel 175mg/m2 IV Q3W if squamous lung cancer
  Other Names: Paclitaxel
Drug: Nab-paclitaxel 260 mg/m2 — nab-paclitaxel 260 mg/m2 Q3W if squamous lung cancer
  Other Names: Nab-paclitaxel

SUMMARY:
To explore the related biomarkers for safety and efficacy of the combination of chemotherapy and tislelizumab in non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and able to understand and agree to comply with study requirements and evaluation forms;
2. Must be at least 18 years of age (or the legal age of commitment in the study occurrence jurisdiction) on the date the informed consent is signed;
3. At least 1 measurable lesion as defined by RECIST v1.1 criteria; Note: Target lesions must be selected to meet one of the following criteria: 1) no prior local therapy or 2) subsequent progression within the previously treated local treatment area as determined by RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Eligible for platinum-based doublet chemotherapy;
6. pre-treatment tumor tissue samples for biomarker analysis can be provided;
7. Adequate hematology and end-organ function as defined by the following laboratory values (≤ 7 days prior to first dose):
8. Patients did not require blood transfusion, platelet transfusion, or growth factor support ≤ 14 days prior to blood draw: i. Absolute neutrophil count ≥ 1.5 * 109/L ii. Platelets ≥ 100 * 109/L iii. Hemoglobin ≥ 90 g/L
9. Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or glomerular filtration rate ≥ 60 mL/min calculated by CKD-EPI formula;
10. AST and ALT ≤ 2.5 times ULN, or AST and ALT ≤ 5 times ULN in patients with a documented history of liver metastases;
11. Serum total bilirubin ≤ 1.5 times ULN (total bilirubin must be < 3 times ULN for patients with Gilbert's syndrome)
12. International normalized ratio (INR) ≤ 1.5 or prothrombin time ≤ 1.5 times ULN;
13. Partial thromboplastin time (APTT) ≤ 1.5 × ULN;
14. Females of childbearing potential must agree to practice highly effective contraception for the duration of the study and for ≥ 120 days after dosing and have a negative serum pregnancy test ≤ 7 days before the first dose of study drug;
15. Nonsterilized men must agree to use highly effective contraception for the duration of the study and for ≥ 120 days after study drug administration;
16. Life expectancy greater than 3 months;

Cohort A Specific Inclusion Criteria:

1. Histologically confirmed Stage IIB-IIIA NSCLC (as defined by the American Joint Committee on Cancer, 8th edition);
2. Confirmed eligibility for R0 resection for curative intent by thoracic surgeon assessment;
3. Adequate cardiopulmonary function, confirmed to meet the requirement for surgical resection for curative intent;

Cohort B Specific Inclusion Criteria:

1) Histologically or cytologically confirmed locally advanced (Stage IIIA-IIIC), or metastatic (Stage IV) NSCLC not amenable to curative surgery or radiotherapy.

Exclusion Criteria:

1. Patients with EGFR mutation, ALK gene rearrangement or ROS1 gene rearrangement:

   1. For patients with non-squamous cell carcinoma, if EGFR mutation status is unknown, tissue samples should be provided for local or central laboratory testing before enrollment;
   2. For patients with squamous cell carcinoma, if EGFR mutation status is unknown, it is not required to conduct test at screening;
   3. Testing at screening is not required if ALK gene rearrangement or ROS1 gene rearrangement status is unknown;
2. Allergic to any study drug or excipients;
3. Patients who have been treated with immune checkpoint inhibitors such as anti-PD-1, PD-L1 or CTLA-4 therapy;
4. Cohort A: patients who have received systemic platinum-based doublet chemotherapy; Cohort B: patients who have received systemic platinum-based doublet chemotherapy as advanced systemic therapy;
5. Patients received other approved systemic anticancer therapy or systemic immunomodulators (including but not limited to interferon, interleukin 2, and tumor necrosis factor) 4 weeks before the first dose;
6. Cohort B: patients with refractory pleural effusion or ascites, such as pleural effusion or ascites requiring puncture and drainage 2 before the first dose;
7. Cohort B: Patients with active leptomeningeal disease or brain metastasis, such as central nervous system symptoms, requiring interventional therapy (including but not limited to radiotherapy, intracranial pressure lowering therapy, etc.);
8. Patients with any disease requiring systemic treatment with corticosteroids (daily dose of prednisone or equivalent > 10 mg) or other immunosuppressive drugs 14 days before grouping; Note: epinephrine replacement steroids (daily dose of prednisone ≤ 10 mg or equivalent) are allowed;Inhaled corticosteroids with minimal intranasal or systemic absorption; prophylactic use of prescription corticosteroids (eg, for contrast medium allergy) for short duration (≤ 7 days) or for treatment of non-autoimmune diseases (eg, delayed hypersensitivity reaction to contact allergens) is permitted;
9. Active autoimmune disease or history of autoimmune disease that may recur; Note: well-controlled type 1 diabetes is allowed; hypothyroidism (controlled with thyroid hormone replacement only); well-controlled celiac disease; skin disease not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia); any other condition that is not expected to recur in the absence of an external trigger.
10. History of interstitial lung disease, pneumonitis or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease;
11. 4. Serious infection occurred before grouping, including but not limited to hospitalization due to infectious complications, bacteremia or severe pneumonia; severe chronic or active infection (including pulmonary tuberculosis infection, etc.) requiring systemic (oral or intravenous) antibiotics within 14 days before grouping;
12. HBV deoxyribonucleic acid (DNA) must be < 500 IU/mL (or 2500 copies/mL) in inactive/asymptomatic carriers, patients with chronic or active hepatitis B virus (HBV) at screening Note: Patients with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should be treated according to treatment guidelines. Patients receiving antiviral therapy at screening should be treated > 2 weeks prior to screening.
13. Any major surgery requiring general anesthesia ≤ 28 before the first dose;
14. Presence of underlying medical conditions or alcohol/drug abuse or dependence that would impair the administration of the study drug, or that could affect the interpretation of the results, or result in a high risk of treatment complications;
15. Simultaneous participation in another therapeutic clinical study;
16. Pregnant or lactating women, or male and female patients planning to have children during the study;
17. Other conditions that the investigators consider inappropriate for participation in this trial, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Drug safety incidents | 90 days after initial treatment of tislelizumab or 30 days post-operation, whichever is later
  Safety as measured by number of participants with Grade 3 and 4 lab abnormalities, as defined by CTCAE v5.0

SECONDARY OUTCOMES:
Evaluation of the major pathologic response (MPR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 36 months
  The major pathologic response is defined as less than 10% tumor cells in the pathologically resected specimen
pathologic complete response | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first，assessed up to 36 months
  defined as no tumor cells observed in pathologically resected specimens
Resectable rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first，assessed up to 36 months
  defined as the number of patients who underwent surgical resection/the number of randomized patients in each group
Disease-free survival | From date of randomization until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60months
  defined as the interval from the surgery to the observation of confirmed disease recurrence

OTHER OUTCOMES:
PD-L1 expression, TMB, and other potential predictive biomarkers, correlated with response to treatment | 36 months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangzhou Medical University Affiliated Cancer Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University cancer center, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangzhou panyu central hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao A, Lin Y, Guan S, Chen Y, Zhai W, Zhou Y, Feng S, Guan Y, Zhang Y, Huang M, Wang X, Long H. Baseline multi-omics signatures could predict therapeutic response to neoadjuvant anti-PD-1 immunochemotherapy in non-small-cell lung cancer. Clin Transl Med. 2026 Jan;16(1):e70579. doi: 10.1002/ctm2.70579. PMID 41499358